CLINICAL TRIAL: NCT04540536
Title: Feasibility and Effectiveness of Real-time, Remote Continuous Glucose Monitoring in Adolescents With Poorly Controlled Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Abha Choudhary, Assistant Professor of Pediatrics, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU-2020-0699
Record Dates: First submitted 2020-07-17; First posted 2020-09-07 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 1; Noncompliance, Patient
Keywords: Type 1 Diabetes; Continuous Glucose Monitors; Telemedicine; Remote Monitoring; Secure Texting; Poorly controlled diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Patient Compliance | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Other: Continuous Glucose Monitoring — Participants will be provided with a Dexcom G6 continuous glucose monitor for the duration of the study.
Other: Secure texting — A secure platform (TigerConnect) will be used for three-way communication between parents, participants, and clinical personnel

SUMMARY:
Adolescents with Type 1 Diabetes (age 13-18 years, T1D duration >6 months managed on insulin) and poor glycemic control will wear a blinded CGM to obtain baseline data. After assuring adherence to CGM wear, participants will receive a non-blinded CGM and will share their blood glucose levels with the study team. Clinical personnel will remotely monitor patients in real-time for 3 months and communicate regularly over secure text messaging with participants and their parents. Following active remote monitoring, the participants will wear a non-blinded CGM for 3 months. Primary outcome assessment will be the change in HbA1c after 3 months of real-time remote continuous glucose monitoring.

ELIGIBILITY:
Inclusion criteria

* Age between 13-18
* Diagnosis of type 1 diabetes for at least six months.
* Both sexes and all ethnicities included.
* Subject and at least one parent able to communicate in English.
* Poorly controlled T1D as evidenced by a >30% annual risk of developing DKA in the following year OR Hemoglobin A1c ≥ 12%
* Treated with subcutaneous insulin, either with a basal/bolus insulin regimen or a continuous subcutaneous insulin infusion (CSII) device.
* Willing to wear CGM and utilize the share function to clinician and guardian, with measuring blood glucose checks as required by the CGM.
* Owning a smartphone compatible with Dexcom G6 software to allow the use of share/follow features with internet access capabilities
* Willing to participate in secure text messaging with study personnel.
* Female participants must have a negative pregnancy test.

Exclusion criteria

* Type 2 diabetes, secondary diabetes or CF related diabetes.
* Other severe chronic disease (e.g., cancer) which in the judgment of the investigator is likely to significantly affect glycemic control.
* Patients cannot be taking systemic corticosteroids at enrollment because of adverse effects on glycemic control, but we will not disqualify subjects who require such therapy during the study. Inhaled or topical corticosteroids are permissible.
* Patients with uncontrolled hypothyroidism (TSH >20) or uncontrolled hyperthyroidism will be excluded from the study. Patients with out of range values may be retested after medication dose adjustment.
* Developmental delay or behavioral disorder in the patient of sufficient severity, in the judgment of the investigator, to interfere with study activities. Severe uncontrolled depression defined as PHQ-9A >15 at time of enrollment is an exclusion criterion.
* Medical or psychiatric disorder in a parent of sufficient severity, in the judgment of the investigator, to interfere with study activities.
* Pregnancy, planned pregnancy or breast feeding
* CGM adhesive allergy
* Skin condition that makes CGM placement contraindicated.
* Sickle cell disease or hemoglobinopathy
* Red blood cell transfusion within 3 months prior to study enrollment

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin A1c after three-month follow-up visit after remote continuous glucose monitoring monitoring and secure text messaging. | 3 months

OTHER OUTCOMES:
Change in depression score after clinical remote CGM monitoring and secure text messaging. | 3 months
  Depression screening will be assessed by Patient Health Questionnaire (PHQ-9A), a depression questionnaire consisting of 9 items answered on a scale from "0" (not at all) to "3" (nearly every day). Total depression severity score ranges of 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Change in quality of life score after clinical remote CGM monitoring and secure text messaging. | 3 months
  Quality of life screening assessed by the Pediatric Quality Life Inventory for teens 13-18, PedsQL4.08, a 23-item questionnaire with a 5-point Likert scale from 0 (never) to 4 (almost always). Items are reversed and then added. The higher the score, the better the quality of life.
Change in self efficacy score after clinical remote CGM monitoring and secure text messaging. | 3 months
  Self-efficacy assessed by The Self-Efficacy for Diabetes Self-Management Measure (SEDM), a 10-item self-report scale that covers the major aspects of diabetes self-management including monitoring blood glucose levels, dosing insulin, food choices, and exercise, and performance of diabetes-related tasks when feeling overwhelmed or frustrated. Total score range for the SEDM is 1-10, with a higher score indicating higher self-efficacy.
Change in parent-child collaboration score after clinical remote CGM monitoring and secure text messaging. | 3 months
  Parent-child collaboration in diabetes care assessed using the Collaborative Parent Involvement Scale, a 12-item questionnaire with a five-point Likert scale, from almost never to always, and is targeted for adolescents. The scale aims to assess parental use of problem solving, teachable moments, diabetes, help with autonomy, and supervision of diabetes care when the adolescent is not around. Higher scores indicate better parent-adolescent collaboration.
Change in depression score 3 months after clinical remote continuous glucose monitoring monitoring and immediately after a period of self-monitoring of CGM data | 6 months
  Depression screening assessed by Patient Health Questionnaire (PHQ-9A), a depression questionnaire consisting of 9 items answered on a scale from "0" (not at all) to "3" (nearly every day). Total depression severity score ranges of 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Change in quality of life score 3 months after clinical remote continuous glucose monitoring monitoring and immediately after a period of self-monitoring of CGM data | 6 months
  Quality of life screening assessed by the Pediatric Quality Life Inventory for teens 13-18, PedsQL4.08, a 23-item questionnaire with a 5-point Likert scale from 0 (never) to 4 (almost always). Items are reversed and then added. The higher the score, the better the quality of life.
Change in self efficacy score 3 months after clinical remote continuous glucose monitoring monitoring and immediately after a period of self-monitoring of CGM data | 6 months
  Self-efficacy assessed by The Self-Efficacy for Diabetes Self-Management Measure (SEDM), a 10-item self-report scale that covers the major aspects of diabetes self-management including monitoring blood glucose levels, dosing insulin, food choices, and exercise, and performance of diabetes-related tasks when feeling overwhelmed or frustrated. Total score range for the SEDM is 1-10, with a higher score indicating higher self-efficacy.
Change in parent-child collaboration score 3 months after clinical remote continuous glucose monitoring monitoring and immediately after a period of self-monitoring of CGM data | 6 months
  Parent-child collaboration in diabetes care assessed using the Collaborative Parent Involvement Scale, a 12-item questionnaire with a five-point Likert scale, from almost never to always, and is targeted for adolescents. The scale aims to assess parental use of problem solving, teachable moments, diabetes, help with autonomy, and supervision of diabetes care when the adolescent is not around. Higher scores indicate better parent-adolescent collaboration.
The percent difference in Hemoglobin A1c after clinical remote monitoring and after self-monitoring of the CGM | 6 months
CGM time in range percentage will be compared between baseline, clinical remote monitoring, and self-monitoring of CGM | 6 months
CGM percent hyperglycemia will be compared between baseline, clinical remote monitoring, and self-monitoring of CGM | 6 months
Mean CGM glucose (in mg/dL) will be compared between baseline, clinical remote monitoring, and self-monitoring of CGM | 6 months
Percent CGM wear will be compared between baseline, clinical remote monitoring, and self-monitoring of CGM | 6 months
Mean time (in minutes) taken for a text to be read by a participant or a guardian. | 3 months
Average time spent by medical provider per participant per day. | 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Childrens Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No